CLINICAL TRIAL: NCT05448703
Title: A Multicenter Prospective Observational Study on Predictive Models and Clinical Outcome of Radiation Pneumonitis
Brief Title: A Study on Predictive Models and Clinical Outcome of Radiation Pneumonitis
Status: Recruiting | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Hubei Cancer Hospital, Tongji Medical College, Huazhong University of Science and Technology (Unknown); Jingjiang People' Hospital (Unknown)
Responsible Party: Principal Investigator, Xianglin Yuan, Professor, Chief Physician, Huazhong University of Science and Technology
Other Study IDs: TJCC012
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Radiation Pneumonitis
MeSH Terms: conditions — Radiation Pneumonitis | interventions — Blood Specimen Collection; Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — From peripheral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Lung cancer patients treated with thoracic radiotherapy
  Interventions: Other: Blood Samples for Biomarkers

INTERVENTIONS:
Other: Blood Samples for Biomarkers — blood sample to be taken at baseline, during radiotherapy, and after radiotherapy

SUMMARY:
Radiation pneumonitis is the main dose-limiting toxicity of thoracic radiotherapy, which can affect life quality, survival, and the tumor-controlling effects of patients receiving thoracic radiotherapy.

The purpose of this study is to:

* Identify biomarkers including serum proteins, gene expression, genetic changes, and epigenetic modifications that determine radiation pneumonitis.
* Investigate the relationship between radiation pneumonitis and other toxicities induced by radiotherapy.
* Construct a predictive model for radiation pneumonitis.
* Evaluate survival and treatment outcome of patients with radiation pneumonitis.

DETAILED DESCRIPTION:
1. Collect clinical information, CT images, and peripheral blood of the lung cancer patients treated with thoracic radiotherapy in Tongji Hospital, Hubei Cancer Hospital, and Jingjiang People's Hospital.
2. Follow up the enrolled patients. All patients enrolled in this study are examined during and one month after radiotherapy. Then, the patients are followed every three months for the first year and every six months thereafter. At each follow-up visits, all patients are asked to undergo a chest CT, and information including survival status, symptoms, CT images, and treatment is collected. Radiation pneumonitis and other toxicities induced by radiotherapy are graded by two radiation oncologists according to the Common Terminology Criteria for Adverse Events 4.0 (CTCAE4.0).
3. Detect serum proteins, gene expression profile, single-nucleotide polymorphisms, and epigenetic modifications that may be associated with radiation pneumonitis.
4. Screen biomarkers that are associated with radiation pneumonitis via univariate and multivariate Cox regression analysis.
5. Construct a predictive model of radiation pneumonitis based on clinical information, radiomics, and biomarkers via machine learning or Least absolute shrinkage and selection operator.
6. Use Kaplan-Meier and Cox model to analyze the association of radiation pneumonitis with survival and efficacy of antitumor treatment.
7. Identify biomarkers and predictors of other toxicities induced by radiotherapy including radiation esophagitis, cardiotoxicity and radiodermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of lung cancer by histology
2. Radiation dose at least 45 Gy
3. Karnofsky >60
4. Age>18
5. Life expectancy of at least 6 months

Exclusion Criteria:

1. Previous thoracic irradiation
2. Severe cardiopulmonary diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients treated with thoracic radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Radiation pneumonitis | 12 months after radiotherapy
  radiation pneumonitis grade >=2 or 3 graded by CTCAE4.0. [Time Frame: 12 months after radiotherapy]
Overall Survival | 5 years after radiotherapy
  A long-term follow up will be scheduled to allow a complete survival analysis.

SECONDARY OUTCOMES:
Other injuries induced by radiotherapy | 5 years after radiotherapy
  Assessment of other common injuries induced by thoracic radiotherapy including injuries in heart, skin, and esophagus according to CTCAE4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xianglin Yuan, PhD, Principal Investigator — Tongji Hospital
Locations (3):
- China (3):
  - Hubei Cancer Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Jingjiang People' Hospital, Jingjiang, Jiangsu